CLINICAL TRIAL: NCT06235190
Title: Assessment of a Novel NeuroAI-powered Transcutaneous Neuromodulation Device in Alleviating Tremor Symptoms and Enhancing Quality of Life for Patients with Upper Limb Essential Tremor
Brief Title: Assessment of the Safety and Efficacy of the Felix NeuroAI Wristband in Essential Tremor
Acronym: TRANQUIL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fasikl Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FSK-CIP-2
Record Dates: First submitted 2024-01-11; First posted 2024-01-31 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 2:1 ratio to Felix and Sham and be followed for 90 days. After the 90-day follow-up, all subjects will be encouraged to participate in the continued access phase, where subjects randomized to the Sham arm will cross over to Felix and all subjects will be followed up to 1 year (from randomization).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Felix NeuroAI Wristband (Experimental)
  Interventions: Device: Felix NeuroAI Wristband
- Sham Device (Sham Comparator)
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: Felix NeuroAI Wristband — The Felix NeuroAI Wristband (Felix) is a wrist-worn, noninvasive, transcutaneous neurostimulation system. Using a proprietary artificial intelligence (AI) algorithm, stimulation will be automatically adapted to patient's needs with the goal to provide full day relief of upper limb tremor.
  Arms: Felix NeuroAI Wristband
Device: Sham Device — The sham device has the same exterior appearance and components as the Felix device and is used the same way (without delivering the treatment).
  Arms: Sham Device

SUMMARY:
The goal of this clinical study is to compare Felix NeuroAI Wristband and sham device in patients with essential tremor. The main question it aims to answer is:

• Is Felix a safe and efficacious treatment for patients with essential tremor?

Participants will be treated with either Felix or Sham for a period of up to 90 days. After that, they will be eligible to participate in a long-term, open-label study and be treated with Felix.

DETAILED DESCRIPTION:
The TRANQUIL study is a prospective, randomized, sham-controlled, double-blinded, multi-center, multi-region trial. The objective of this clinical investigation is to evaluate the safety and effectiveness of the Felix NeuroAI Wristband to aid in the relief of upper limb tremor in adults with essential tremor (ET).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Willing to provide written, informed consent to participate in the study.
* A clinical diagnosis of ET by a movement disorder specialist.
* For the dominant hand, a tremor severity score of 2 or higher as measured by one of the TETRAS Performance Subscale (PS) tasks (items 4, 6, 7, and 8) and a total score of 7 or higher across these items. If applicable, this must be met while the patient is on ET treatment.
* Stable dosage of anti-tremor medications, if applicable, for 30 days prior to study entry.
* Stable dosage of antidepressant medications, if applicable, for 90 days prior to study entry.
* Familiar with operating a touch-screen smartphone and connecting to Wi-Fi internet at home.
* If necessary, have a dedicated caregiver to help with study required activities, such as putting on the study device, etc.
* Willing to comply with study protocol requirements including:

  1. Remaining on a stable dosage of anti-tremor and antidepressant medications, if applicable, during the course of the study.
  2. Do not start any new anti-tremor treatment during the course of the study (except the assigned treatment in the study).
  3. Remaining on stable caffeine consumption, if applicable, during the course of the study.
  4. No alcohol or marijuana consumption the day before a study visit.
  5. Do not share study/device-related information on the internet or with other study patients.

Exclusion Criteria:

* Prior limb amputation or any known symptomatic peripheral neuropathy condition of the involved upper extremity.
* Prior surgical intervention for ET such as deep brain stimulation or thalamotomy.
* Moderate to severe alcohol use disorder (AUD) as per Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) (the presence of at least 4 symptoms or more).
* Any current drug abuse.
* Use of recreational drugs other than marijuana.
* Current unstable epileptic conditions with a seizure within 6 months of study entry.
* Other possible causes of tremor such as drug-induced tremor, enhanced physiological tremor, dystonia, and Parkinson's disease.
* Pregnant or nursing subjects and those who plan pregnancy during the course of the study.
* Swollen, infected, inflamed areas, or skin eruptions, open wounds, or cancerous lesions of skin at the stimulation site.
* Known allergy to adhesive bandages.
* The presence of any cognitive or other impairment that in the judgement of the investigator will impede the assessment of study outcomes.
* Botulinum Toxin injection for hand tremor within 4 months prior to study enrollment.
* History of use of other transcutaneous afferent patterned stimulation (TAPS) devices such as Cala Trio.
* Subject is currently participating or has participated in another interventional clinical trial in the last 30 days which may confound the results of this study, unless approved by the Sponsor.
* Subject is unable to communicate with the investigator and study staff.
* Any health condition that in the investigator's opinion should preclude participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in Tremor Research Group Essential Tremor Rating Assessment Scale (TETRAS) modified Activities of Daily Living (mADL) score from baseline pre-stimulation to Day 90 | 90 days
  TETRAS mADL score is a composite sum of items 2 to 11 of the TETRAS ADL subscale and items 6 (bilateral) and 7 (dominant hand) of the TETRAS performance subscale (PS). Each item is scored from 0 to 4, indicating increasing severity of tremor. TETRAS mADL score is calculated as the sum of all 12 items and ranges from 0 to 52.

SECONDARY OUTCOMES:
Change in Tremor Research Group Essential Tremor Rating Assessment Scale (TETRAS) modified Activities of Daily Living (mADL) score from baseline pre-stimulation to 14 days, 30 days, 60 days, 180 days, and 1 year | 14 days, 30 days, and 60 days, 180 days, and 1 year
  TETRAS mADL score is a composite sum of items 2 to 11 of the TETRAS ADL subscale and items 6 (bilateral) and 7 (dominant hand) of the TETRAS performance subscale (PS). Each item is scored from 0 to 4, indicating increasing severity of tremor. TETRAS mADL score is calculated as the sum of all 12 items and ranges from 0 to 52.
Responder Rate | 14 days, 30 days, 60 days, 90 days, 180 days, and 1 year.
  Responder rate is defined as the proportion of patients responding to the treatment, as defined by change in TETRAS mADL score at or above a pre-specified margin.
Tremor Research Group Essential Tremor Rating Assessment Scale (TETRAS) performance subscale (PS) Items 1, 4, and 8 | Baseline, 30 days, 90 days, and 1 year
  Each TETRAS PS item is scored by physician from 0 to 4, indicating increasing severity of tremor.
Tremor Research Group Essential Tremor Rating Assessment Scale (TETRAS) performance subscale (PS) Items 6 and 7 | Baseline,14 days, 30 days, 60 days, 90 days, 180 days, and 1 year.
  Each TETRAS PS item is scored by physician from 0 to 4, indicating increasing severity of tremor.
Tremor Research Group Essential Tremor Rating Assessment Scale (TETRAS) performance subscale (PS) Dominant Hand Score | Baseline, 30 days, 90 days, and 1 year
  The sum of TETRAS PS items 4, 6, 7, and 8 for the dominant hand. Each item is scored by physician from 0 to 4, indicating increasing severity of tremor.
Clinical Global Impression of Severity (CGI-S) | Baseline, 30 days, 90 days, and 1 year
  Physician rating on a 7-point scale, from 1 (normal) to 7 (amongst the most extreme tremor)
Patient Global Impression of Severity (PGI-S) | Baseline, 14 days, 30 days, 60 days, 90 days, 180 days, and 1 year.
  Patient rating on a 7-point scale, from 1 (normal) to 7 (amongst the most extreme tremor)
Clinical Global Impression of Improvement (CGI-I) | Baseline, 30 days, 90 days, and 1 year
  Physician rating of tremor improvement on a 7-point scale, from 1 (very much improved) to 7 (very much worse)
Patient Global Impression of Improvement (PGI-I) | Baseline, 14 days, 30 days, 60 days, 90 days, 180 days, and 1 year.
  Patient rating of tremor improvement on a 7-point scale, from 1 (very much improved) to 7 (very much worse)
Quality of Life in Essential Tremor Questionnaire (QUEST) | Baseline, 90 days, and 1 year
  QUEST is a 30-item scale developed specifically for patients with essential tremor to measure items impacting perceived quality of life (QOL) that generic QOL measures do not effectively capture, including activities of daily living that are affected by essential tremor.
Tremor power | Continuously measured up to 1 year
  Device measured tremor power. Unit: (m/s^2)^2
Patient survey | 14 days, 30 days, 60 days, 90 days, 180 days, and 1 year
  Patient survey of satisfaction with the treatment and the durability of the treatment effect

CONTACTS AND LOCATIONS:
Locations (12):
- United States (8):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Parkinson's Research Centers of America - Palo Alto, Palo Alto, California
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - The University Of Kansas Medical Center, Kansas City, Kansas
  - Parkinson's Research Centers of America - Long Island, Commack, New York
  - Columbia University Irving Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Houston Methodist Research Institute, Houston, Texas
- China (4):
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Xuanwu Hospital Capital Medical University, Beijing
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Derived] Ondo WG, Lv W, Zhu X, Hu Y, Isaacson SH, Yuan Y, Espay AJ, Kreitzman D, Kuo SH, Brillman S, Shill HA, Lyons KE, Yang Z, Zhao Q, Zhang Z, Pahwa R. Transcutaneous Peripheral Nerve Stimulation for Essential Tremor: A Randomized Clinical Trial. JAMA Neurol. 2025 Dec 1;82(12):1235-1242. doi: 10.1001/jamaneurol.2025.3905. PMID 41114984